CLINICAL TRIAL: NCT05776316
Title: Culturally Response Integrated Harm Reduction Services for Black and Latinx People Who Use Drugs
Brief Title: Harm Reduction Services
Acronym: HRS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 22-01089
Record Dates: First submitted 2023-03-06; First posted 2023-03-20 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Drug Use; Substance Abuse; Mental Illness
Keywords: Harm Reduction; Latinx/Hispanix; Black/African American; Drug Use; Cocaine; Opioids; Methamphetamines
MeSH Terms: conditions — Substance-Related Disorders; Mental Disorders; Harm Reduction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IHRI (Experimental): Integrated harm reduction intervention (IHRI) program tailored specifically for highly marginalized Black and Latinx people who use drugs (PWUDs). The IHRI lasts 8 weeks in duration, with the first 4 weeks consisting of weekly education lessons provided by the IHRI care coordinator. The subsequent 4 weeks will involve individualized identification of vulnerabilities in the social determinants of health (SDOH) for the purposes of making informed referrals to relevant partnering social service organizations. Participants will also be exposed to service encounters through mobile vans in which staff offer information to PWUD on syringe exchange, clean user kits, naloxone use, and fentanyl strip distribution.
  Interventions: Behavioral: Integrated Harm Reduction Intervention (IHRI)
- HR SAU (No Intervention): Harm reduction services as usual (HR SAU). Participants will be exposed to service encounters through the mobile vans in which staff offer information to PWUD on syringe exchange, clean user kits, naloxone use, and fentanyl strip distribution.

INTERVENTIONS:
Behavioral: Integrated Harm Reduction Intervention (IHRI) — 8-week program targeting areas rooted in the 8 principles of harm reduction. Includes weekly education lessons and informed referrals to social service organizations.
  Arms: IHRI

SUMMARY:
The purpose of this study is to assess whether an integrated harm reduction intervention (IHRI), compared to harm reduction (HR) services as usual, will improve harm reduction service utilization among Black and Latinx people who use drugs (PWUD).

ELIGIBILITY:
Inclusion Criteria:

* at least 18 years of age
* self-identified as misusing opioids +/- other substances (stimulants) in the past 30 days, confirmed by interview using DSM-5 criteria
* English or Spanish speaking
* able to provide informed consent.

Exclusion Criteria:

* inability to provide informed consent or participate in the study procedures as proposed in the consent
* active suicidal or homicidal ideation or an unstable psychotic disorder (schizophrenia, schizoaffective disorder) or mood disorder (bipolar disorder, severe major depressive disorder)
* an unwillingness to be randomized.
* are prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-11-26 (Actual); Primary Completion 2026-03-27 (Estimated); Study Completion 2028-03-28 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants who Attend At least 1 Harm Reduction (HR) Session after Introductory HR Session | Up to Week 8
  Measure of engagement.
Percentage of Participants who Attend at least 3 HR Sessions in Total | Up to Week 8
  Measure of engagement.

SECONDARY OUTCOMES:
Change from Baseline in Number of Days of Opioid/Other Stimulant Use | Baseline, Week 8
  Number of days of opioid/other stimulant use will be calculated using the timeline follow back method, which asks participants to estimate how many days over the previous 30 days that they used opioids/other stimulants.
Change from Baseline in Overdose Risk Assessment Tool Score | Baseline, Week 8
  20-item assessment of overdose risk. Each item prompts a "Yes" or "No" response. If the response is "Yes," a score is assigned for that item. If the answer is "No," no score is assigned for that item. The total score is the sum of responses and ranges from 0 to 42; lower scores indicate low risk, higher scores indicate higher risk. A decrease in scores indicates risk of overdose decreased during the observatioN period.
Change from Baseline in Brief Quality of Life Scale Score | Baseline, Week 8
  12-item assessment of quality of life. Each item is ranked on a 5-point Likert scale ranging from 0 (do not agree at all) to 4 (agree completely). The total score is the sum of responses and ranges from 0 to 48; higher scores indicate higher quality of life. An increase in scores indicates quality of life increased during the observation period.

CONTACTS AND LOCATIONS:
Overall Officials: Ayana Jordan, MD, PhD, Principal Investigator — NYU Langone Health
Locations (3):
- United States (3):
  - Yale University, New Haven, Connecticut
  - NYU Langone Health, New York, New York
  - Nathan Kline Institute, Orangeburg, New York

IPD SHARING:
Plan to Share IPD: Yes
The de-identified participant data collected during the trial will be shared upon reasonable request beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research provided the investigator who proposes to use the data executes a data use agreement with NYU Langone Health. Requests may be directed to: [Ayana.Jordan@nyulangone.org]. The protocol, statistical analysis plan, informed consent form, and clinical study report will be made available on Clinicaltrials.gov.
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: Researchers who provide a methodologically sound proposal, as well as investigators whose proposed use of the data has been approved by an independent review committee ("learned intermediary") identified for this purpose, will be granted access to achieve the aims in the approved proposal. Requests should be directed to Ayana.Jordan@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.